CLINICAL TRIAL: NCT03941860
Title: Optimizing Prolonged Treatment In Myeloma Using MRD Assessment (OPTIMUM)
Brief Title: Testing the Addition of Ixazomib/Placebo to Lenalidomide in Patients With Evidence of Residual Multiple Myeloma, OPTIMUM Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2019-02790; NCI-2019-02790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAA171 (Other: ECOG-ACRIN Cancer Research Group); EAA171 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Fluid Therapy; Biopsy; ixazomib; Lenalidomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (lenalidomide, ixazomib citrate) (Experimental): Patients receive lenalidomide PO QD on days 1-28 and ixazomib citrate PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspirate and/or biopsy and PET and CT scan at screening and on study as well as undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ixazomib Citrate; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (lenalidomide, placebo) (Placebo Comparator): Patients receive lenalidomide PO QD on days 1-28 and a placebo PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspirate and/or biopsy and PET and CT scan at screening and on study as well as undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Lenalidomide; Other: Placebo Administration; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow aspirate
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN 9708; MLN-9708; MLN9708; Ninlaro
  Arms: Arm A (lenalidomide, ixazomib citrate)
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Other: Placebo Administration — Given PO
  Arms: Arm B (lenalidomide, placebo)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Arm B (lenalidomide, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well lenalidomide in combination with ixazomib works compared to lenalidomide alone in treating patients with evidence of residual multiple myeloma after stem cell transplantation. Lenalidomide may help shrink or slow the growth of multiple myeloma. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving lenalidomide and ixazomib together may work better than giving lenalidomide alone in treating patients with evidence of residual multiple myeloma after a stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether escalating maintenance therapy with the addition of ixazomib citrate (ixazomib) to lenalidomide improves overall survival (OS) among patients who are minimal residual disease (MRD) positive after approximately 1 year of lenalidomide maintenance following an early stem cell transplant (=< 12 months from diagnosis).

SECONDARY OBJECTIVES:

I. To establish whether progression-free survival (PFS) is superior with the addition of ixazomib to lenalidomide maintenance.

II. To evaluate best response on treatment and compare response rates between arms.

III. To evaluate the safety profile of ixazomib added to lenalidomide and compare toxicity rates between arms.

EXPLORATORY OBJECTIVES:

I. To measure treatment exposure and adherence. II. To estimate treatment duration, duration of response and time to progression.

PATIENT-REPORTED OUTCOMES (PRO) OBJECTIVES:

I. To quantify the extent to which the addition of ixazomib to lenalidomide maintenance contributes to neuropathy and associated physical and functional impairments. (Primary) II. To assess the impact of the addition of ixazomib to lenalidomide maintenance on disease control and associated physical and functional well-being. (Primary) III. To evaluate time to worsening and recovery rate related to neuropathy. (Secondary) IV. To evaluate time to improvement and response rate related to disease control. (Secondary) V. To evaluate attributes of select patient reported treatment-emergent symptomatic adverse events (Patient-Reported Outcomes - Common Terminology Criteria for Adverse Events [PRO-CTCAE]) longitudinally and compare responses with provider-reported adverse events. (Exploratory) VI. To measure the likelihood of medication adherence and examine the relationship with treatment exposure. (Exploratory) VII. To assess correlation among patient reported outcome measures and association with clinical outcomes. (Exploratory) VIII. To tabulate PRO compliance and completion rates. (Exploratory)

IMAGING OBJECTIVES:

I. To evaluate the association between baseline fludeoxyglucose F-18 (18F-FDG)-positron emission tomography (PET)/computed tomography (CT) and patient outcomes.

II. To compare overall survival (OS) with the addition of ixazomib to lenalidomide among baseline 18F-FDG PET/CT-positive and 18F-FDG PET/CT -negative subgroups.

III. To compare the change in quantitative 18F-FDG PET/CT parameters over time with the addition of ixazomib to lenalidomide.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-28 and ixazomib citrate PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspirate and/or biopsy and positron emission tomography (PET) and computed tomography (CT) scan at screening and on study as well as undergo collection of blood samples throughout the trial.

ARM B: Patients receive lenalidomide PO QD on days 1-28 and a placebo PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspirate and/or biopsy and PET and CT scan at screening and on study as well as undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 3 months if < 2 years from study entry, every 6 months if 2-5 years from study entry, then every 12 months for up to 10 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: PRE-REGISTRATION
* Patient must be >= 18 years of age
* Patient must be previously diagnosed with multiple myeloma (MM) and be on lenalidomide maintenance with >= 5mg daily for at least 6 months and no more than 18 months after an early autologous stem cell transplantation (SCT =< 12 months of diagnosis). Patient must not be off lenalidomide maintenance therapy for more than 30 days prior to start of treatment on Step 1 of this protocol
* Patient must be able to undergo a diagnostic bone marrow aspirate following pre-registration to Step 0

  * NOTE: A bone marrow aspirate specimen must be submitted to Mayo Clinic Hematology Laboratory for central assessment of minimal residual disease (MRD) status to confirm patient's eligibility for Step 1 randomization. Mayo Clinic will forward results to the submitting institution within three (3) business days of receipt of the bone marrow specimen
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Patient must have been able to maintain at least 5mg daily dose of lenalidomide without growth factor support
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* STEP 1 RANDOMIZATION
* Patient must meet Step 0 eligibility criteria at the time of Step 1 randomization
* Patients must have evidence of residual disease by central MRD testing or by presence of monoclonal protein in serum or urine
* Patient must have serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), and serum free light chain (FLC) performed =< 28 days prior to randomization

  * NOTE: UPEP (on a 24-hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hour (hr). Please note that if both serum and urine M-components are present, both must be followed in order to evaluate response
* Hemoglobin >= 8 g/dL (obtained =< 14 days prior to randomization)
* Untransfused platelet count >= 75,000 cells/mm^3 (obtained =< 14 days prior to randomization)
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3 (obtained =< 14 days prior to randomization)
* Calculated creatinine clearance >= 30 mL/min (obtained =< 14 days prior to randomization)
* Total bilirubin =< 1.5 times the upper limit of normal (ULN) (obtained =< 14 days prior to randomization)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 times the upper limit of normal (ULN) (obtained =< 14 days prior to randomization)
* Patient must agree to register into the mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) registered trademark program and be willing and able to comply with the requirements of Revlimid REMS registered trademark
* Patients of childbearing potential must either abstain from sexual intercourse for the duration of their participation in the study or agree to use TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME for 1) at least 28 days before starting study treatment; 2) while participating in the study; 3) during dose interruptions; and 4) for at least 90 days after the last dose of protocol treatment. Patients must also agree to not breastfeed during this same time period. Men must agree to either abstain from sexual intercourse for the duration of their participation in the study or use a latex condom during sexual contact with a partner of childbearing potential while participating in the study and for 90 days after the last dose of protocol treatment even if they have had a successful vasectomy. Patients must also agree to abstain from donating sperm while on study treatment and for 28 days after the last dose of protocol treatment even if they have had a successful vasectomy. All patients must agree to abstain from donating blood during study participation and for at least 28 days after the last dose of protocol treatment

Exclusion Criteria:

* Patient must not have primary refractory or progressive disease on a proteasome inhibitor-based regimen during induction therapy prior to stem cell transplant
* Patient must not be on other concurrent chemotherapy, or any ancillary therapy considered investigational

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy and are allowed while on protocol treatment
* Patient must not have uncontrolled psychiatric illness or social situations that would limit compliance with study requirements
* Patient must not have another malignancy requiring treatment or have received treatment within two years before pre-registration or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patients must not have known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or lenalidomide including difficulty swallowing
* Patient must not have known hepatitis B surface antigen-positive status or known or suspected active hepatitis C infection, but testing specifically for the trial is not required
* Patient must not be off lenalidomide maintenance therapy for more than 30 days prior to start of treatment on Step 1 of this protocol
* Patients must not have grade 2 or higher peripheral neuropathy or grade 1 peripheral neuropathy with pain per Common Terminology Criteria for Adverse Events (CTCAE)
* Patients must not have uncontrolled intercurrent illness
* Patients must not have grade 2 or higher diarrhea per CTCAE in the absence of antidiarrheals
* Patients must not have been on systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (such as rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort
* Patient must not be pregnant due to potential harm to the fetus from ixazomib and lenalidomide. All patients of childbearing potential must have a blood test or urine study with a sensitivity of at least 25 mIU/mL within 10-14 days prior to the first dose of lenalidomide and again within 24 hours prior to the first dose of lenalidomide. Patients of childbearing potential must also agree to ongoing pregnancy testing while on treatment. A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K Kumar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (222):
- United States (221):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on June 1, 2021 and closed to accrual on March 3, 2023 due to slow accrual.
Period: Overall Study
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data is not reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months if patient is <2 years from randomization, every 6 months if patient is 2-5 years from randomization, annually if patient is 5 years or more from randomization.
Population: Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data is not reported.
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival defined as the time from randomization until the earlier of progression or death due to any cause, or censored at date of last disease evaluation.
  Progression is defined as one of the following criteria is met.
  * Increase of ≥ 25% from lowest value reported in serum M-component (the absolute increase must be ≥ 0.5 g/dL) and/or urine M-component (the absolute increase must be ≥ 200 mg/ 24 hours).
  * Only in patients without measurable serum and urine M protein levels: the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL.
  * If the only measurable disease is bone marrow, bone marrow plasma cell percentage: the absolute % must be ≥ 10%.
  * Development of new bone lesions or soft tissue plasmacytomas or ≥ 50% increase from nadir in the size (SPD) of existing bone lesions or soft tissue plasmacytoma or ≥ 50% increase in the longest diameter of a previous lesion > 1cm in short axis.
Time Frame: as for outcome 1
Population: Only one patient was enrolled on this study. Due to confidentiality reasons, individual data was not reported.
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Best Response on Treatment
Description: Response is evaluated based on standard International Myeloma Working Group (IMWG) criteria and tabulated by category. Response (stringent complete response [sCR], complete response [CR], very good partial response [VGPR]) is defined as below.
  sCR: All CR criteria and the following have to be met. Normal serum FLC ratio at two consecutive times and absence of clonal cells in bone marrow by immunohistochemistry or 2- to 4- color flow cytometry. Presence/absence of clonal cells is based upon the κ/λ ratio. An abnormal κ/λ ratio by immunohistochemistry requires a minimum of 100 plasma cells for analysis. An abnormal ratio reflecting presence of an abnormal clone is κ/λ ratio of 4:1 or 1:2.
  CR: Complete disappearance of an Mprotein and no evidence of myeloma in the bone marrow.
  VGPR: Serum M-protein detectable by immunofixation but not quantifiable on electrophoresis and urine M-protein < 100 mg/24 hours
Time Frame: as for outcome 1
Population: Only one patient was enrolled on this study. Due to confidentiality reasons, individual data was not reported.
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo)
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Cumulative Dose
Description: Cumulative dose will be calculated as the sum of all doses taken across all cycles.
Time Frame: End of treatment, up to 10 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Relative Dose Intensity
Description: Relative dose intensity will be calculated as the dose intensity divided by planned dose intensity.
Time Frame: End of treatment, up to 10 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Dose Intensity
Description: Will be calculated as cumulative dose received divided by treatment duration. Will be calculated overall and by cycle. Data will be summarized by treatment arm with descriptive statistics and graphically over time.
Time Frame: Up to 15 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Treatment Duration
Description: Treatment duration is defined as the time from randomization to date off treatment. Patients who are still on treatment will be censored at the date of last treatment.
Time Frame: End of treatment, up to 10 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Duration of Response
Description: Duration of response is defined as the time from observed response (VGPR, CR or sCR) to the time of progression in the respective group of responders.
Time Frame: as for outcome 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time to Progression
Description: Time to progression is defined as the time from randomization to progression. Patients without documented progression will be censored at date of last disease assessment.
  Progression is defined as one of the following criteria is met.
  * Increase of ≥ 25% from lowest value reported in serum M-component (the absolute increase must be ≥ 0.5 g/dL) and/or urine M-component (the absolute increase must be ≥ 200 mg/ 24 hours).
  * Only in patients without measurable serum and urine M protein levels: the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL.
  * If the only measurable disease is bone marrow, bone marrow plasma cell percentage: the absolute % must be ≥ 10%.
  * Development of new bone lesions or soft tissue plasmacytomas or ≥ 50% increase from nadir in the size (SPD) of existing bone lesions or soft tissue plasmacytoma or ≥ 50% increase in the longest diameter of a previous lesion > 1cm in short axis.
Time Frame: as for outcome 1
Reporting Status: Not Posted

10. Other Pre Specified Outcome: To Determine the Extent and Timing of Neuropathy Associated With the Addition of Ixazomib to Lenalidomide Maintenance on Patient Reported Health-related Quality of Life (QOL) Outcomes.
Description: Health-related QOL will be assessed with three instruments: 1) the FACT-General (G) functional well-being (FWB) and physical wellbeing (PWB) subscales. Each FACT-G subscale has 7 items. The 14 items are based on a 5-point Likert scale (0-4) resulting in a score ranging from 0 to 56 points with a higher score indicating better health-related QOL; 2) The FACT/GOG-Neurotoxicity Trial Outcomes Index (FACT/GOG-Ntx TOI) comprised of the FWB and PWB subscales plus the neurotoxicity subscale which has 11 items, summing to a score of 0-100; and 3) the FACT-Multiple Myeloma Trial Outcomes Index (FACT-MM TOI) comprised of the FWB and PWB subscales plus the multiple myeloma subscale which has 14 items, summing to a score of 0-112 for the instrument.
Time Frame: Assessed at baseline, end of every 3 cycles for the first 24 cycles, every 6 cycles thereafter up to completion of 48 cycles, and at treatment discontinuation prior to completing 48 cycles. During long-term follow-up, 4 quarterly assessments for 1 year.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: To Assess the Impact and Timing of Disease Control With the Addition of Ixazomib to Lenalidomide Maintenance on Patient Reported Healthrelated Quality of Life Outcomes
Description: as for outcome 10
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Presence, Frequency, Interference, Amount, and/or Severity of Select Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: NCI PRO-CTCAE items will be administered. There are 80 symptomatic AE terms included in the PRO-CTCAE library. Items correspond to 5 attributes measured [frequency (F), severity (S), interference (I), presence/absence (P) and amount (A)] based on multiple choice questions. Response for each attribute except P which is binary is on a 5-point Likert scale with 5 indicating 'almost constantly' frequency, 'very severe' severity, 'very much' amount or 'very much' interference. For each attribute, recall is the past 7 days. Attributes measured for each symptomatic AE varies and comprise the PRO-CTCAE item library. For this study, 23 symptomatic AEs summing to 38 items have been selected as presented below. There are 10 symptomatic AEs assessed using one item, 11 symptomatic AEs assessed using two items, and 6 symptomatic AEs assessed using three items. The types of items in order of prevalence include severity, interference, frequency, present/not present, and amount. T
Time Frame: Assessed every cycle up to cycle 25
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Adherence Starts With Knowledge (ASK)-12 Scores
Description: The Adherence Starts with Knowledge Scale (ASK-12) will be used to assess the likelihood that a patient is taking oral medications per protocol. The 12-item questionnaire was derived from the predecessor ASK-20 using a study population of 112 patients with asthma, congestive heart failure or diabetes. In this study, the ASK12 had good internal consistency, and test-retest reliability. The ASK-12 which elicits the same type of information as the Morisky Medication Adherence Scale (MMAS) also demonstrated convergent validity through strong correlation with MMAS-4 (Spearman correlation r = 0.74; p < 0.001). The ASK-12 titled 'Taking Medicine What Gets in the Way?' is segmented into 3 sections: inconvenience/forgetfulness (3 items), treatment beliefs (4 items) and behavior (5 items). Response for each item is on a 5-point Likert scale (1-5) with the total score ranging from 12-60 and a higher score representing less likelihood of medication adherence.
Time Frame: Assessed at cycles 7, 13, 19, 25, 31, 37, 43 and 49
Reporting Status: Not Posted

14. Other Pre Specified Outcome: To Assess Correlation Among Patient Reported Outcome Measures and Association With Clinical Outcomes.
Description: The association between patient reported outcome measures and clinical outcomes will be evaluated.
Time Frame: as for outcome 1
Reporting Status: Not Posted

15. Other Pre Specified Outcome: PRO Compliance Rate
Description: PRO compliance rate is defined as the proportion of patients who submit the given PRO instrument among those eligible at each time point which excludes those missing by design (due to death or disease progression, early treatment discontinuation).
Time Frame: At 10 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: PRO Completion Rate
Description: PRO completion rate is defined as the proportion of patients who complete given PRO instrument based on the instrument's scoring system among those eligible at each time point.
Time Frame: Assessed at each cycle, up to 10 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: To Evaluate the Association Between Baseline 18F-FDG PET/CT and Patient Outcomes.
Description: Quantitatively, the association between baseline standardized uptake values (SUV) based quantitative 18F-FDG PET/CT parameters (SUVmax, SUVpeak, metabolic tumor volume [MTV], total lesion glycolysis [TLG]) and PFS will be analyzed through Cox regression. PFS will be defined as the time from randomization until the earlier of progression or death due to any cause. SUV-based quantitative 18F-FDG PET/CT (qPET) parameters will be analyzed as continuous covariates.
Time Frame: as for outcome 1
Reporting Status: Not Posted

18. Other Pre Specified Outcome: To Compare the Change in Quantitative 18F-FDG PET/CT Parameters Over Time With the Addition of Ixazomib to Lenalidomide
Description: The difference in qPET parameters from the baseline 18FFDG PET/CT to the year 1 18F-FDG PET/CT will be reported by study arm. An analysis of covariance (ANCOVA) model will be used to test for a treatment effect on each qPET parameter, where the baseline qPET parameter value and an indicator for study arm are included as covariates, with the qPET parameter at year 1 as the model outcome.
Time Frame: Assessed at baseline and 1 year
Reporting Status: Not Posted

19. Other Pre Specified Outcome: To Compare Overall Survival (OS) With the Addition of Ixazomib to Lenalidomide Among Baseline 18F-FDG PET/CT-positive and 18F-FDG PET/CT-negative Subgroups.
Description: Heterogeneity of treatment effect will be assessed at full information, using a two-sided statistical test for interaction between study arm (ixazomib/lenalidomide vs. placebo/lenalidomide) and baseline 18F-FDG PET/CT status (positive/abnormal vs. negative) in a Cox regression model. If the statistical test for interaction is not significant at the 0.05 level, we will conclude that there is not sufficient evidence for heterogeneity of treatment effect; if the statistical test for interaction is significant, estimated treatment hazard ratios for OS (ixazomib arm vs. placebo arm) will be reported separately for baseline 18FFDG PET/CT-positive and 18F-FDG PET/CT-negative subgroups, along with the corresponding 95% confidence intervals. OS will be defined as the time from randomization until death or the date last known alive.
Time Frame: as for outcome 1
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Incidence of Adverse Events
Description: Incidence of adverse events
Time Frame: Assessed at each cycle, up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks until 30 days after treatment completion, up to 10 years
Description: Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data is not reported.
Arm/Group | Arm A (Lenalidomide, Ixazomib Citrate) | Arm B (Lenalidomide, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data is not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03941860/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03941860/ICF_001.pdf